CLINICAL TRIAL: NCT01081977
Title: Effect of Timing of Umbilical Cord Clamping on Haematological and Clinical Outcomes of Infants at Birth and Three Months of Age
Brief Title: Effect of Timing of Umbilical Cord Clamping on Haematological and Clinical Outcomes of Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor and Founding Chair, Division of Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 991-Ped/ERC-08
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Anemia; Ferritin; Complications; Hemorrhage; Jaundice
Keywords: Delayed cord clamping; Ferritin; Hemoglobin; Neonatal anemia; Postpartum haemorrhage; Neonatal jaundice
MeSH Terms: conditions — Anemia; Hemorrhage; Jaundice; Anemia, Neonatal; Postpartum Hemorrhage; Jaundice, Neonatal | interventions — Umbilical Cord Clamping; Ferritins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Cord Clamping Group (Active Comparator): Early Cord Clamping Group (Clamping of Umbilical Cord within 30 seconds of shoulder delivery of neonate).
  Interventions: Procedure: Early Cord Clamping
- Delayed Cord Clapming Group (Experimental): Delayed Umbilical Cord Clamping Group (Clamping of Umbilical Cord within 2 minutes of shoulder delivery of neonate).
  Interventions: Procedure: Delayed Cord Clamping

INTERVENTIONS:
Procedure: Early Cord Clamping — Early Umbilical Cord Clamping (Clamping of Umbilical Cord within 30 seconds of shoulder delivery of neonate)
  Other Names: Cord clamping; Neonate; Anemia
  Arms: Early Cord Clamping Group
Procedure: Delayed Cord Clamping — Delayed Umbilical Cord Clamping (Clamping Umbilical Cord after 2 minutes of shoulder delivery of neonate
  Other Names: Cord clamping; Ferritin; Infant
  Arms: Delayed Cord Clapming Group

SUMMARY:
In developing countries up to 50% of children become anemic by 12 months of age(1. Iron deficiency anemia is a major risk factor for neonatal and infantile mortality and morbidity in Pakistan. It has detrimental effects on neurodevelopment of infants and may be irreversible even after iron therapy(2). Type of cost effective interventions during perinatal period for prevention of anemia in later infancy is limited. Delayed cord clamping has a beneficial effect on prevention of anemia in later infancy because of increased iron stores at birth(3. However there are controversies in incorporating delayed cord clamping practice in the management of third stage of labour globally(4) Paucity of national guidelines and lack of substantial data in Pakistan on this topic strongly necessitates such study trials. This study may contribute to develop a protocol on the timing of cord clamping which will be cost effective in prevention of iron deficiency anemia in the investigators infantile population.

The investigators will conduct a randomized controlled trial and the investigators hypothesis is that delayed cord clamping will result in higher hemoglobin (Hb), hematocrit (Hct) and ferritin at third month as compared to early cord clamping.

OBJECTIVES:

A- Primary:

1. To study the effect of timing of umbilical cord clamping on hemoglobin (Hb), Hematocrit (Hct) at birth, 48 hours and Hb, Hct and ferritin at three months of age.
2. To study the effect of timing of umbilical cord clamping on short term clinical profile of neonates like jaundice, respiratory distress, anemia, polycythemia etc. during fist 24 to 48 hours of life.

B- Secondary:

To assess whether delayed cord clamping is associated with undesirable effects on mothers followed till 48 hours postpartum.

DETAILED DESCRIPTION:
Delayed umbilical cord clamping (DCC) results in approximately 30-40 ml additional placental blood volume transfusion to the neonate and 30-35 mg increase in iron stores at birth(5).The neonatal benefits include higher hematocrit (Hct), higher red blood cells flow to vital organs, better cardiopulmonary adaptation, additional iron stores and less anemia in later infancy(6).It is evident from different studies that no adverse effects of DCC have been noticed in mothers as well as in their neonates(7). The beneficial effect of delayed cord clamping is not only observed in term infants but it has a positive impact on preterm and small for gestational age (SGA) infants too. The requirement of packed cell transfusion in first six months has significantly reduced as noticed from different studies(8).It is also associated with lower risk of intraventricular hemorrhage and late onset sepsis in preterm infants(9).

The practice of early cord clamping (ECC) is commonly following in our maternity units. It is believed that it reduces the risk of post partum haemorrhage (PPH) and duration of third stage of labour. But at the same time it does not provide any benefit to the neonate(4).Conversely it increases the possibility of fetomaternal transfusion, hypovolemic damage, neonatal anemia, respiratory distress syndrome and type 2 diabetes in later life(5).The risk of iso immunization in rhesus negative mothers are also increased with ECC(10).

ELIGIBILITY:
Inclusion Criteria:

* Mother-infant pairs, between 35 weeks and 41 completed weeks of pregnancy, planned to deliver through vaginal or Elective lower segment cesarean section(ELSCS)

Exclusion Criteria:

* Women with multiple gestation
* Complications like pregnancy induced hypertension (PIH), Gestational diabetes Mellitus (GDM), Pre/Eclampsia, placental insufficiency, suboptimal CTG (late deceleration, variable deceleration)
* Rh-isoimmunization
* Chronic maternal illnesses (hypertension, cardiomyopathies, chronic renal diseases, haemoglobinopathies
* Pre-existing risk factor for postpartum haemorrhage, like polyhydramnios, previous PPH
* Infants with antenatal diagnosis of congenital malformations of any system (CVS, GIT, RENAL CNS ,RESP), anomalies or syndromes
* Emergency caesarean section (EmLSCS)
* Need for neonatal resuscitation at birth and NICU admission due to causes not directly related to the intervention trial.

Criteria 1 to 6 will be applied before randomization and criteria 7 and 8 assess after randomization.

Ages: 1 Minute to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Hematological Characteristics of Infants | From Birth to Third month of age
  Infantile hematological characteristics ( hemoglobin, hematocrit at birth(cord),48 hours of age and Hemoglobin, Hematocrit and serum ferritin at third month).
Short term Clinical Profiles | From birth to 48 hours of age
  Short term neonatal clinical profile (respiratory distress, polycythemia hematocrit ≥65%), neonatal anemia , clinical jaundice hyperbilirubinemia),requirement of phototherapy or exchange transfusion)

SECONDARY OUTCOMES:
Maternal Characteristics | From Delivery to 48 hours postpartum
  Maternal characteristics ( Primary PPH, duration of third stage of labour ≥ 30 min, mean blood loss during the third stage of labour, need for therapeutic oxytocin, manual removal of placenta and Hb at 48 hours postpartum).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Zulfiqar Bhutta, MBBS, PhD, Study Director — Aga Khan University; Dr Huma Shaireen, MBBS, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] 1. World Health Organozation. Newborns: No longer going unnoticed. The World Health Report:2005.p 79-101. . 2005 [updated 2005; cited]; Available from: http://www.who.int/whr/2005/en/. 2. Shafir T, Angulo-Barroso R, Jing Y, Angelilli ML, Jacobson SW, Lozoff B. Iron deficiency and infant motor development. Early Hum Dev. 2008 Jul;84(7):479-85. 3. Hutton EK, Hassan ES. Late vs early clamping of the umbilical cord in full-term neonates: systematic review and meta-analysis of controlled trials. JAMA. 2007 Mar 21;297(11):1241-52. 4. Ononeze AB, Hutchon DJ. Attitude of obstetricians towards delayed cord clamping: a questionnaire-based study. J Obstet Gynaecol. 2009 Apr;29(3):223-4. 5. Bhutta ZA, Ahmed T, Black RE, Cousens S, Dewey K, Giugliani E, et al. What works? Interventions for maternal and child undernutrition and survival. Lancet. 2008 Feb 2;371(9610):417-40. 6. Zaramella P, Freato F, Quaresima V, Secchieri S, Milan A, Grisafi D, et al. Early versus late cord clamping: effects on peripheral blood flow and cardiac function in term infants. Early Hum Dev. 2008 Mar;84(3):195-200. 7. McDonald SJ, Middleton P. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2008(2):CD004074. 8. Strauss RG, Mock DM, Johnson KJ, Cress GA, Burmeister LF, Zimmerman MB, et al. A randomized clinical trial comparing immediate versus delayed clamping of the umbilical cord in preterm infants: short-term clinical and laboratory endpoints. Transfusion. 2008 Apr;48(4):658-65. 9. Mercer JS, Vohr BR, McGrath MM, Padbury JF, Wallach M, Oh W. Delayed cord clamping in very preterm infants reduces the incidence of intraventricular hemorrhage and late-onset sepsis: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):1235-42. 10. Levy T, Blickstein I. Timing of cord clamping revisited. J Perinat Med. 2006;34(4):293-7.